CLINICAL TRIAL: NCT06102980
Title: Estimation of Liver Fibrosis in Patients With MASLD Screening Criteria Through Endoscopic Ultrasound-guided Shear Wave vs Transabdominal Ultrasound and Transient Elastography: The RUMIPAMBA Diagnostic Trial
Brief Title: Endoscopic Ultrasound Shear Wave for Liver Fibrosis in MASLD Patients: The RUMIPAMBA Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Principal Investigator, Carlos Robles-Medranda, Head of the Endoscopy Division, Instituto Ecuatoriano de Enfermedades Digestivas
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IECED-02102023
Record Dates: First submitted 2023-10-02; First posted 2023-10-26 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Liver Steatosis; Fibrosis, Liver
Keywords: Liver steatosis; Fatty liver; Endosonography; Elastography; Liver fibrosis
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis | interventions — Endosonography

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: After EUS-SWE, a clinical research coordinator will open the label to confirm the patient's cohort. The patient will undergo the EUS-guided two-lobe liver biopsy only if the patient belongs to the liver steatosis group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MASLD screening patients (Active Comparator): Patients with requirements of screening following the European Association for the Study of the Liver (EASL) 2016 recommendations. The MASLD screening group will be compounded by patients with at least one of the following criteria:
  1. Over fifty years old;
  2. Body mass index (BMI) over 25 kg/m2;
  3. Diabetes mellitus type 2;
  4. Metabolic syndrome; or
  5. Persistently elevated liver enzymes.
  Interventions: Device: Transparietal ultrasound (US)-based shear wave elastography (SWE) attenuation measurement; Device: Transparietal ultrasound (US)-based shear wave elastography (SWE) stiffness measurement; Device: Vibration-controlled transient elastography (VCTE) attenuation measurement; Device: Vibration-controlled transient elastography (VCTE) stiffness measurement; Device: Endoscopic ultrasound (EUS)-guided shear wave elastography (SWE) stiffness measurement
- Controls (Other): Patients without requirements of screening following the European Association for the Study of the Liver (EASL) 2016 recommendations. The control group will be compounded by patients who will not present any of the following criteria:
  1. Over fifty years old;
  2. Body mass index (BMI) over 25 kg/m2;
  3. Diabetes mellitus type 2;
  4. Metabolic syndrome; and
  5. Persistently elevated liver enzymes.
  To be a control participant does not mean that the patient is a healthy participant. The control participants are patients who request any type of endoscopy and fulfil the criteria not to screen for liver steatosis. For example, a 48-year-old male with 21 kg/m2 BMI, without diabetes mellitus type 2, any metabolic syndrome-related comorbidities, with normal liver enzymes and who refused an episode of persistently elevated liver enzymes, with persistent reflux disease after two months of proton pump inhibitor therapy,
  Interventions: Device: Transparietal ultrasound (US)-based shear wave elastography (SWE) attenuation measurement; Device: Transparietal ultrasound (US)-based shear wave elastography (SWE) stiffness measurement; Device: Vibration-controlled transient elastography (VCTE) attenuation measurement; Device: Vibration-controlled transient elastography (VCTE) stiffness measurement; Device: Endoscopic ultrasound (EUS)-guided shear wave elastography (SWE) stiffness measurement

INTERVENTIONS:
Device: Transparietal ultrasound (US)-based shear wave elastography (SWE) attenuation measurement — The operator will be blinded to any clinical record. Before US-SWE, the patient must be fasted for a minimum of 4 hours and must remain alcohol-free for 7 days. Using an Aloka Arietta 850 (Olympus America, PA, USA), each patient must be supine. Upon breath-hold at the end of expiration, ten measurements will be obtained with the probe placed in the area of the right hepatic lobe through an intercostal space.
  Other Names: US-SWE attenuation
Device: Transparietal ultrasound (US)-based shear wave elastography (SWE) stiffness measurement — The operator will be blinded to any clinical record. Before US-SWE, the patient must be fasted for a minimum of 4 hours and must remain alcohol-free for 7 days. Using an Aloka Arietta 850 (Olympus America, PA, USA), each patient must be supine. Upon breath-hold at the end of expiration, ten measurements will be obtained with the probe placed in the area of the right hepatic lobe through an intercostal space.
  Other Names: US-SWE stiffness
Device: Vibration-controlled transient elastography (VCTE) attenuation measurement — The operator will be blinded to any clinical record. Before VCTE, the patient must be fasted for a minimum of 4 hours and must remain alcohol-free for 7 days. Using the FibroScan® Compact 530 (Echosens, Paris, France), each patient must be supine with the right arm in abduction and the ipsilateral hand resting under the head. Upon breath-hold at the end of expiration, ten measurements will be obtained with the M-probe placed in the area of the right hepatic lobe through an intercostal space. Transition to an extra large probe will be based on a VCTE automatic probe selection tool prompt.
  Other Names: VCTE attenuation
Device: Vibration-controlled transient elastography (VCTE) stiffness measurement — The operator will be blinded to any clinical record. Before VCTE, the patient must be fasted for a minimum of 4 hours and must remain alcohol-free for 7 days. Using the FibroScan® Compact 530 (Echosens, Paris, France), each patient must be supine with the right arm in abduction and the ipsilateral hand resting under the head. Upon breath-hold at the end of expiration, ten measurements will be obtained with the M-probe placed in the area of the right hepatic lobe through an intercostal space. Transition to an extra large probe will be based on a VCTE automatic probe selection tool prompt.
  Other Names: VCTE measurement
Device: Endoscopic ultrasound (EUS)-guided shear wave elastography (SWE) stiffness measurement — EUS-SWE will be performed by an experienced endoscopist, blinded to clinical records. The expert will use the ArrietaTM 850 EUS console (Fujifilm, Tokyo, Japan) using a linear ultrasound video gastroscope EUS-J10 (Pentax Medical, Hoya Corp, Japan). Both lobes will be evaluated. The transducer will be positioned in the gastric window to visualize right liver segment number five and left liver segment two or three. The elastogram region of interest (ROI) will be placed within the liver tissue at a distance ≥10 mm beneath the hepatic capsule in an area free of vessels and artefacts. A 10-mm circular ROI will be placed within the elastogram at a depth of 4-5 cm from the skin, and a minimum of ten successful kilopascal measurements will be obtained.
  In the first stage of this research, the EUS-SWE measurement will be limited to the estimation of liver fibrosis only. Currently, available EUS-SWE equipment does not allow the estimation of the attenuation.
  Other Names: EUS-SWE attenuation

SUMMARY:
Currently, there is no description of the contribution of the endoscopic ultrasound (EUS)-guided shear wave elastography (SWE) when describing liver fibrosis in patients with screening criteria of metabolic dysfunction-associated steatotic liver disease (MASLD), with absent-to-mild liver fibrosis. Similar research has been published but using vibration-controlled transient elastography (VCTE), recommended mainly due to its lower cost and less invasiveness. However, VCTE is limited to the anatomical proportions of the patient's body, and cannot assess the right hepatic lobe with less reliability, contrary to the EUS-SWE.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD), formerly non-alcoholic fatty liver disease (NAFLD), is an umbrella term which involves simple liver steatosis, metabolic-associated steatohepatitis (MASH) and MASH-related liver cirrhosis. Liver steatosis relies on imaging or biomarkers, but liver biopsy remains the gold standard for its diagnosis and grading. It comprehends intracellular accumulation of triacylglycerol (TAG) as microvascular or macrovascular lipid droplets in at least 5% of hepatocytes. Liver biopsy is invasive, requires a high-quality biopsy sample, can mislead a diagnosis due to sampling bias, depends on pathologist interpretation variability and implies adverse events related to the punction.

There are non-invasive resources useful for the screening and surveillance of liver steatosis and fibrosis. Apart from serum biomarkers, non-invasive technologies designed for this purpose use transabdominal ultrasound (US)-based elastography, namely: US strain, acoustic radiation force impulse (ARFI), point shear wave elastography (pSWE), two-dimension shear wave elastography (2D-SWE) and vibration-controlled transient elastography (VCTE). Although VCTE presents anatomical limitations when used in overweight patients or assessing the right hepatic lobe, it is largely accepted by international guidelines for assessing liver steatosis and fibrosis. Endoscopic ultrasound (EUS)-guided shear wave elastography (SWE) is independent of the anatomical proportions of the patients, and it permits a more reliable right hepatic lobe evaluation. However, it is an invasive and high-cost procedure.

VCTE, US-ARFI and EUS-SWE determine liver fibrosis quantitatively in terms of liver stiffness through kiloPascals. There are four important gaps in the literature: First, the diagnostic accuracy of VCTE for liver steatosis has been profoundly analysed in NAFLD, but in a wide spectrum of liver fibrosis patients, from absent to cirrhosis. These limits finding extrapolations for screening and surveillance. Second, comparisons between VCTE, US-ARFI and EUS-SWE have concentrated on liver fibrosis or cirrhosis, but they have not been compared head-to-head in the context of absent-to-mild liver fibrosis vs controls. Third, there is no determined diagnostic accuracy for EUS-SWE for an early liver fibrosis estimation in MASLD patients. It is useful considering EUS is becoming a more popular procedure. Finally, and to be consequent with the third point, the identification and grading of liver steatosis and fibrosis still need to be described in the nowadays called MASLD patients.

The present study aims to determine the difference in the estimation of liver fibrosis among VCTE, US-ARFI and EUS-SWE in patients with clinical criteria of MASLD screening but absent-to-mild liver fibrosis, according to non-invasive methods.

This study has been called by the authors through the acronym RUMIPAMBA, which means "Role of endoscopic Ultrasound-guided shear wave for MASLD-related liver steatosis and fibrosis Identification in Patients with Absent to Mild Basal fibrosis, based on non-invasive Analytical laboratory tests". In the general culture, Rumipamba is the name of an archaeological prehispanic and preincaic park from Quito, the capital city of Ecuador.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for any kind of endoscopic procedure.
* Without clinical suspicion of advanced liver fibrosis.
* Acceptance to participate in the study.

Exclusion Criteria:

* History of greater amounts of alcohol per week (140 g/week and 210 g/week for females and males respectively).
* Significant or advanced fibrosis by Fibrosis-4 Index (FIB4) or the aspartate aminotransferase to platelet ratio index (APRI).
* Any liver space-occupying lesion in the US.
* Comorbidities or conditions related to avoidance of interventional procedures, namely: pregnancy or nursing, coagulopathy or any risk of bleeding, Anaesthesiology Society Association classification IV or higher, New York Heart Association functional class III or IV.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Vibration-controlled transient elastography (VCTE) liver steatosis grade | Six months
  Liver steatosis will be defined by elastography using the controlled attenuation parameter (CAP), measured in decibels per meter.
Transparietal ultrasound (US)-based shear wave elastography (SWE) liver steatosis grade | Six months
  Liver steatosis will be defined by elastography using the attenuation coefficient (ATT), measured in decibels per meter. The ATT corresponds to the VCTE CAP measurement.
Endoscopic ultrasound (EUS)-guided shear wave elastography (SWE) liver steatosis grade | Six months
  Liver steatosis per hepatic lobe will be defined by elastography using the attenuation coefficient (ATT) measurement. The ATT corresponds to the VCTE CAP measurement.
Endoscopic ultrasound (EUS)-guided liver biopsy steatosis grade | Six months
  The EUS-guided liver biopsy findings, per hepatic lobe, will be standardised through the steatosis-Activity-Fibrosis (SAF) score. The SAF scores steatosis (0-3), ballooning degeneration (0-2), lobular inflammation (0-2), and fibrosis (0-4). Liver steatosis is present when proper steatosis is present, and when both features of activity (ballooning and lobular inflammation) display at least grade 1.

SECONDARY OUTCOMES:
Vibration-controlled transient elastography (VCTE) liver fibrosis grade | Six months
  Liver steatosis will be defined by elastography using kilopascals.
Transparietal ultrasound (US)-based shear wave elastography (SWE) liver fibrosis grade | Six months
  Liver steatosis will be defined by elastography using kilopascals.
Endoscopic ultrasound (EUS)-guided shear wave elastography (SWE) liver fibrosis grade | Six months
  Liver steatosis per hepatic lobe will be defined by elastography using kilopascals.
Endoscopic ultrasound (EUS)-guided liver biopsy fibrosis grade | Six months
  The EUS-guided liver biopsy findings, per hepatic lobe, will be standardised through the Brunt system.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas (IECED)
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas (IECED) Gastroclinica SA, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yazdani L, Rafati I, Gesnik M, Nicolet F, Chayer B, Gilbert G, Volniansky A, Olivie D, Giard JM, Sebastiani G, Nguyen BN, Tang A, Cloutier G. Ultrasound Shear Wave Attenuation Imaging for Grading Liver Steatosis in Volunteers and Patients With Non-alcoholic Fatty Liver Disease: A Pilot Study. Ultrasound Med Biol. 2023 Oct;49(10):2264-2272. doi: 10.1016/j.ultrasmedbio.2023.06.020. Epub 2023 Jul 21. PMID 37482477
- [Background] Liu GT, Ni QF, Zhang YH, Dong XM, Zhou C, Shen B, Zhu JY, Chen YJ, Zhu Z. Application of noninvasive test (acoustic attenuation imaging and ultrasonic shear wave elastography) to grade nonalcoholic fatty liver disease: An observational study. Medicine (Baltimore). 2023 Aug 11;102(32):e34550. doi: 10.1097/MD.0000000000034550. PMID 37565905
- [Background] De A, Duseja A. Natural History of Simple Steatosis or Nonalcoholic Fatty Liver. J Clin Exp Hepatol. 2020 May-Jun;10(3):255-262. doi: 10.1016/j.jceh.2019.09.005. Epub 2019 Sep 20. PMID 32405182
- [Background] Pandyarajan V, Gish RG, Alkhouri N, Noureddin M. Screening for Nonalcoholic Fatty Liver Disease in the Primary Care Clinic. Gastroenterol Hepatol (N Y). 2019 Jul;15(7):357-365. PMID 31391806
- [Background] Kohli DR, Mettman D, Andraws N, Haer E, Porter J, Ulusurac O, Ullery S, Desai M, Siddiqui MS, Sharma P. Comparative accuracy of endosonographic shear wave elastography and transcutaneous liver stiffness measurement: a pilot study. Gastrointest Endosc. 2023 Jan;97(1):35-41.e1. doi: 10.1016/j.gie.2022.08.035. Epub 2022 Aug 29. PMID 36049537